CLINICAL TRIAL: NCT06547528
Title: An Open-label, Uncontrolled, Phase I Dose Escalation Study to Investigate the Tolerability and Safety of ONO-4685 Given as Monotherapy in Patients With Relapsed or Refractory T Cell Lymphoma and Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Brief Title: A Phase I Study to Investigate the Tolerability and Safety of ONO-4685 Given as Monotherapy in T Cell Lymphoma and CLL/SLL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4685-05
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Relapsed or Refractory T Cell Lymphoma and Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ONO-4685 (Experimental)
  Interventions: Drug: ONO-4685

INTERVENTIONS:
Drug: ONO-4685 — ONO-4685 is administered by IV infusion. The administration of ONO-4685 will be continued until disease progression or unacceptable toxicity is observed.

SUMMARY:
A Phase I Study to Investigate the Tolerability and Safety of ONO-4685 Given as Monotherapy in T Cell Lymphoma and CLL/SLL

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histopathologically confirmed diagnosis of one of the following subtypes as defined by the 2017 revision of the WHO classification of lymphoid malignancies:

   Peripheral T-cell lymphoma(PTCL)
   * Angioimmunoblastic T-cell lymphoma(AITL)
   * Peripheral T-cell lymphoma, NOS(PTCL-NOS)
   * Nodal peripheral T-cell lymphoma with TFH phenotype(nodal PTCL with TFH)
   * Follicular T-cell lymphoma(FTCL) Cutaneous T-cell lymphoma(CTCL)
   * Mycosis fungoides(MF)
   * Sezary syndrome Chronic lymphocytic leukemia/small lymphocytic lymphoma(CLL/SLL)
2. Relapsed or refractory patients with tumors for which no established standard therapy is available, or refractory or intolerant to existing standard therapy judged by principal investigator or subinvestigator
3. ECOG PS 0~2
4. Life expectancy of at least 3 months

Exclusion Criteria:

1. Patients with severe complications.
2. Patients with multiple cancers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities(DLT) | Up to 3 Weeks
Incidence and severity of AEs and SAEs | Through study completion, an average of 1 year
Laboratory abnormality profile of ONO-4685 as measured by incidence and severity of clinical laboratory abnormalities | Through study completion, an average of 1 year
Body temperature | Through study completion, an average of 1 year
Pulse rate | Through study completion, an average of 1 year
Systolic/diastolic blood pressure | Through study completion, an average of 1 year
Change of weight during the trial period | Through study completion, an average of 1 year
Chest X-ray test | Through study completion, an average of 1 year
ECG parameters by 12 lead ECG(pulse rate) | Through study completion, an average of 1 year
ECG parameters by 12 lead ECG(RR) | Through study completion, an average of 1 year
ECG parameters by 12 lead ECG(QT interval) | Through study completion, an average of 1 year
ECG parameters by 12 lead ECG(corrected QT intervals [QTcF, QTcB]) | Through study completion, an average of 1 year
ECG parameters by 12 lead ECG(PR interval) | Through study completion, an average of 1 year
ECG parameters by 12 lead ECG(QRS) | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Best overall response (BOR) | Through study completion, an average of 1 year
Overall response rate (ORR) | Through study completion, an average of 1 year
Complete response rate (CRR) | Through study completion, an average of 1 year
Duration of response (DOR) | Through study completion, an average of 1 year
Progression Free Survival(PFS) | Through study completion, an average of 1 year
Time to response (TTR) | Through study completion, an average of 1 year
Overall Survival(OS) | Through study completion, an average of 1 year
The percent change of tumor volume | Through study completion, an average of 1 year
Pharmacokinetics(Cmax) | Through study completion, an average of 1 year
Pharmacokinetics(Tmax) | Through study completion, an average of 1 year
Pharmacokinetics(AUC) | Through study completion, an average of 1 year
Pharmacokinetics(Ceoi) | Through study completion, an average of 1 year
Pharmacokinetics(T1/2) | Through study completion, an average of 1 year
Pharmacokinetics(Ctrough) | Through study completion, an average of 1 year
Volume of distribution(Vd) | Through study completion, an average of 1 year
clearance(CL) | Through study completion, an average of 1 year
Anti-ONO-4685 antibody | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (14):
- Japan (14):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Akita University Hospital, Akita, Akita
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Tokai University Hospital, Isehara-shi, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kindai University Hospital, Osaka Sayama-shi, Osaka
  - Osaka University Hospital, Osaka-fu, Osaka
  - Cancer Institute Hospital of JFCR, Koto-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No